CLINICAL TRIAL: NCT02770144
Title: The Impact of Family Financial Support on Child Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Adam Schickedanz, Clinical Instructor in Pediatrics and Clinical Scholar, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UCLASchickedanzFCCH
Record Dates: First submitted 2016-03-25; First posted 2016-05-12 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Child Overall Health Related Quality of Life
Keywords: Child Quality of Life; Financial Coaching; Socioeconomic Status; Social Determinants of Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Financial Coaching & Social Services Referral (Experimental): Enrollment in one-to-one financial coaching intervention to support savings, income, and credit while reducing debt using available tools in the community development field.
  Interventions: Behavioral: Financial Coaching; Behavioral: Access to Referral to Social Services
- Access to Referrals to Social Services (Active Comparator): Enrollment provides access to referrals to social services to meet basic needs.
  Interventions: Behavioral: Access to Referral to Social Services

INTERVENTIONS:
Behavioral: Financial Coaching — Enrollment in one-to-one financial coaching intervention to support savings, income, and credit while reducing debt using available tools in the community development field.
  Arms: Financial Coaching & Social Services Referral
Behavioral: Access to Referral to Social Services

SUMMARY:
The investigators have partnered with financial coaching organizations to establish what the investigators have termed a "Medical-Financial Partnership (MFP)" that offers financial coaching to improve financial and mental health.The investigators will evaluate the MFP's impact on child overall health rating.

DETAILED DESCRIPTION:
Financial coaching is a new tool in the field of community development, but it has already demonstrated significant financial impact in a number of studies, including one randomized trial conducted by the Urban Institute. Financial coaching improves participant financial literacy, budgeting, saving for financial emergencies, and debt level. The investigators' project will help clinicians and the field of community economic development understand health and well-being through a new economic lens and assess the health-related impacts of the emerging field of financial coaching. The investigators have partnered with financial coaching organizations to establish what they have termed a "Medical-Financial Partnership (MFP)" that offers financial coaching to improve financial and mental health. The investigators will evaluate the MFP's impact on parent-rated child overall health on a 5 point likert scale (Excellent to Poor).

Community-based participants will be recruited from South Los Angeles and randomized to receive either monthly financial coaching plus access to referral for social services (intervention) or access to referral for social services alone (control). Inclusion criteria include having dependents under age 18, having some form of income, and having a tax identification number (social security number or Individual Tax Identification Number). Participants will be surveyed quarterly regarding their parent-rated child overall health on a 5 point likert scale (Excellent to Poor).

ELIGIBILITY:
Inclusion Criteria:

* Participants will include caregivers and parents with one or more dependent children, some form of income, and a tax identification number.

Exclusion Criteria:

* Inability to take part in financial coaching or primary language other than English or Spanish.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-03; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Parent-Rated Child Overall Health | Up to One Year
  Parent-rated overall child health (Excellent, Very Good, Good, Fair, Poor) assessed using a single-item questionnaire. The single item used to assess this outcome is the first item in the Patient Reported Outcomes Measurement Information System child health related quality of life questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Schickedanz, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- LIFT-LA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Participant consent does not include data sharing beyond the study and there is no appropriate repository for such data.